CLINICAL TRIAL: NCT02243332
Title: Dynamic Quadriceps Muscle Stimulation for Treatment of Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Articulate Labs (Industry)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALI-KS-001
Record Dates: First submitted 2014-09-12; First posted 2014-09-17 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Patellofemoral Pain Syndrome; Anterior Knee Pain Syndrome
Keywords: Knee; Pain; Joint; Rehabilitation; Patellofemoral Pain Syndrome; Anterior Knee Pain Syndrome; Knee Pain; Quadriceps
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device (rehabilitation assistance) (Experimental): Device: KneeStim mobile rehabilitation assistance device
  Interventions: Device: KneeStim mobile rehabilitation assistance device

INTERVENTIONS:
Device: KneeStim mobile rehabilitation assistance device — KneeStim is a neuromuscular electrical stimulation (NMES) device that integrates motion-tracking hardware like three-axis accelerometers and a real-time operating system to enable quadriceps muscle stimulation in time with user gait. It is a completely non-invasive device that looks like a light brace and fastens to the user's quadriceps and gastrocnemius muscles. The end goal of this device is to assist with muscle re-strengthening and re-education during a user's everyday activities.
  Other Names: KneeStim

SUMMARY:
The purpose of this small, pilot study is to evaluate a novel device that uses neuromuscular electrical stimulation to assist quadriceps muscles as a user walks. This study will involve use of this device on individuals with patellofemoral pain, a relatively common injury among active people, to see if quadriceps stimulation could mitigate disparities in quadriceps activation timing that may indirectly lead to knee pain.

DETAILED DESCRIPTION:
The interventional device will be tested with 20 women aged 18-40 with evidence of patellofemoral pain syndrome (PFPS) and without any co-morbidities that would confound data or contraindications for NMES use. All participants will be enrolled at a single site (Developmental Motor Lab at the University of Texas), and all of a single participant's testing will be complete within a single day with no requirement for follow-up or long-term participation. Participants will have their gait and quadriceps muscle activation patterns evaluated through four six-minute walk tests (6MWT). The first 6MWT will be without a device, second with a device worn but not activated, third with a device activated and stimulating quadriceps musculature, and the fourth without a device.

Primary Objective: The purpose of this study is to investigate whether electrical stimulation of the vastus medalis (VM) and/or vastus lateralis (VL) to establish coactivation of these muscles during terminal swing phase impacts severity of PFPS symptoms

Secondary Objectives: Secondary purposes for this study include evaluating KneeStim and seeing if there is any evidence of proof of concept in two main areas:

KneeStim as a therapeutic device that may assist individuals with joint rehabilitation KneeStim's on-board operating system and motion tracking system as an effective way to monitor joint kinematics.

This pilot study has a prospective, controlled, single-center design. Participants and investigators will not be blinded to the treatment. Individuals who evaluate the motion-tracking data between VICON and KneeStim will not be informed which data set aligns with which treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40 years
* Symptomatic PFPS on Patella Glide Test, Patella Tilt Test, and Patellar Apprehension Test.

Exclusion Criteria:

* Rheumatoid arthritis or inflammatory arthritis as assessed by licensed physician
* Use of walking aids other than a cane more than 50% of the time in ambulation
* Diagnosed knee disorder other than patellofemoral syndrome
* Pacemaker use, unstable angina, or decompensated heart failure
* Knee replaced in preceding 12 months or replacement planned within 6 months
* Moderate to severe dementia
* Pregnancy (self report)
* Altered sensation at the knee such that the patient is unable to perceive the presence of pinprick.
* Use of intra-articular viscosupplementation or steroid injection within preceding 2 months.
* Use of chronic anticoagulation medication.
* Movement-limiting pain in the back, hip, ankle, or foot of either lower limb.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Measured Quadriceps Musculature Co-Contraction | 20, 40, 60, 80 minutes from start of single-day testing
  Electromyographic (EMG) readings of vastus lateralis and vastus medialis contraction patterns will be taken after four six-minute walk tests (6MWTs) to evaluate any short-term changes in co-contraction.
  6MWT #1: Without interventional device being worn; 6MWT #2: With interventional device being worn, but unpowered; 6MWT #3: With interventional device being worn and operational; 6MWT #4: Without interventional device being worn
  The time period in which a partipant will be involved is not expected to exceed 90 minutes.

SECONDARY OUTCOMES:
Anterior Knee Pain | 20, 40, 60, 80 minutes from start of single-day testing
  Measured with Anterior Knee Pain Scale (AKPS) after each Six Minute Walk Test.
Device Joint Model Accuracy | 20, 40, 60, 80 minutes from start of single-day testing
  The interventional device uses an on-board operating system that determines stimulation timing and location based on modeled joint kinematics. Movement data will be taken from the device and evaluated against movement data measured by a VICON motion-tracking system during each six-minute walk test to evaluate the accuracy of the device's modeled joint kinematics.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Griffin, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- Developmental Motor Control Lab; University of Texas at Austin, Austin, Texas, United States